CLINICAL TRIAL: NCT05916781
Title: Effectiveness of Mycophenolate Mofetil Combined With Tacrolimus for Steroid Tapering in Systemic Lupus Erythematosus: A Prospective, Random Control, Open-label, Single Center Clinical Trial
Brief Title: Effectiveness of Mycophenolate Mofetil Combined With Tacrolimus for Steroid Tapering in Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR008
Record Dates: First submitted 2023-06-09; First posted 2023-06-23 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: mycophenolate mofetil; tacrolimus; steroid tapering; systemic lupus erythematosus; lupus nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Mycophenolic Acid; Tacrolimus; Glucocorticoids

STUDY DESIGN:
Intervention Model Description: First, participants are randomly assigned into 2 groups: steroid tapering group and steroid maintenance group. In steroid tapering group, participants without flare will be assigned into 2 groups: mycophenolate mofetil group and tacrolimus group. In steroid maintenance group, participants without flare will stop the use of steroid for 6 months. Participants without lupus flare after the stop of steroid will be assigned into 2 groups: mycophenolate mofetil group and tacrolimus group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid tapering group (Experimental): 0~6th month: mycophenolate mofetil (1g/d) + tacrolimus (2.0mg/d) + steroid (1 pill/d) 6th~18th month: mycophenolate mofetil (1g/d) + tacrolimus (2.0mg/d) 18th~30th month: Participants who stop steroid treatment and do not flare will be randomly assigned to monotherapy with mycophenolate mofetil or tacrolimus
  Interventions: Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Glucocorticoid
- steroid maintenance group (Active Comparator): 0~18th month: mycophenolate mofetil (1g/d) + tacrolimus (2.0mg/d) + steroid (1 pill/d) 18th~24th month: Participants who do not flare will stop the use of steroid. 24th~30th month: Participants who do not flare will be randomly assigned to monotherapy with mycophenolate mofetil or tacrolimus
  Interventions: Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Glucocorticoid

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Participants in steroid tapering group will take MMF+TAC during the first 18 months. After 18 months, participants without lupus flare will randomly stop MMF or TAC.
  Participants in steroid maintenance group will take MMF+TAC during the first 24 months. After 24 months, participants without lupus flare will randomly stop MMF or TAC.
  Other Names: MMF
Drug: Tacrolimus — Participants in steroid tapering group will take MMF+TAC during the first 18 months. After 18 months, participants without lupus flare will randomly stop MMF or TAC.
  Participants in steroid maintenance group will take MMF+TAC during the first 24 months. After 24 months, participants without lupus flare will randomly stop MMF or TAC.
  Other Names: TAC
Drug: Glucocorticoid — Participants in steroid tapering group will stop taking glucocorticoid after the first 6 months.
  Participants in steroid maintenance group will consistently take glucocorticoid for 18 months, and stop the use of glucocorticoid after 18 months if they do not flare.

SUMMARY:
The goal of this clinical trial is to determine whether mycophenolate mofetil(MMF) combined with tacrolimus(TAC) can maintain remission in patients with lupus nephritis (LN) who have reached treatment targets after steroid tapering. The main question[s] it aims to answer are:

* The efficacy, safety and tolerability of MMF combined with TAC regimen in the treatment of LN patients in the maintenance period.
* The influence of low-dose steroid on carotid intima thickness (CIMT).
* The omics and cell-free RNA (cfRNA) spectral differences related to lupus flare.
* The differences in health economics between steroid tapering and steroid maintenance patients.

Participants will be randomly assigned into 2 groups. In the steroid tapering group, participants will take MMF+TAC treatment without steroid for 1 year, and participants who stop steroid treatment without lupus flare will be randomly assigned to monotherapy with MMF or TAC. In the steroid maintenance group, participants will take MMF+TAC+steroid for 1 year, and participants without lupus flare will stop the use of steroid for 6 months. Participants without lupus flare after the stop of steroid will be randomly assigned to monotherapy with MMF or TAC.

DETAILED DESCRIPTION:
According to the references, with the maintenance of steroid, 1-year lupus flare rate is 7%. Investigators plan to take a 2-year follow-up for participants, so the proportion of patients without flare in steroid maintenance group should be 86%. As this is a non-inferiority study, investigators hypothesize that in steroid tapering group, the proportion of patients without flare is also 86%. Investigators set α=0.05 (two-sided), 1-β=0.90, non-inferiority value = 15%, the dropout rate = 20%. The sample size of each group should be 110, the 220 in total.

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus participants diagnosed with 2019 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria, fulfilled with American College of Rheumatology (ACR) lupus nephritis definition, and have reached treatment target (accord with lupus nephritis clinical remission and DORIS) for at least 6 months. The target is defined as: (1)24h urine protein ≤0.5g/d；(2)stable of improved renal function (baseline creatinine ±10% or decrease 15%)；(3)clinical SLE Disease Activity Index (cSLEDAI) =0 (all scores are required zero, except hypocomplementemia and anti-dsDNA antibody positivity)；(4)PGA score (Physician Global Assessment)<0.5; (5)prednisone or equivalent steroid dose≤5mg/d；(6)stable use of immunosuppressants and antimalarial drugs; (7)no use of biological agents.
* According to the physician, the participant can accept this treatment.
* The participant is willing to join this clinical trial, has good compliance, and could understand and sign the informed consent before the study begins.

Exclusion Criteria:

* SLE complicated with important organ dysfunction, including consciousness disorder, cognitive disorder, renal dysfunction, heart dysfunction (NYHA class 3, 4), pulmonary arterial hypertension, and interstitial lung disease.
* SLE with active vital organ disease (not satisfied with DORIS), including but not limited to active neuropsychiatric systemic lupus erythematosus, lupus nephritis, thrombocytopenia, hemolytic anemia, myocardial involvement, gastrointestinal involvement, etc.
* Participants who are allergic to or intolerant with mycophenolate mofetil or tacrolimus.
* Participants with acute and chronic infections requiring anti-infective treatment, including but not limited to tuberculosis infection, Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infection, Human Immunodeficiency Virus (HIV) infection, and Cytomegalovirus (CMV) infection.
* Participants who are pregnant or planning to become pregnant.
* Participants who have used biological agents within 6 months before enrollment.
* The researcher considers any condition that may cause the participant to be unable to complete the study or bring an obvious risk to the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The 1-year flare rate of lupus nephritis participants who reach the treatment target and accept MMF+TAC remedy tapering steroid in the maintenance period. | 6th~18th month
  If the DORIS (Definition of Remission In SLE) is not sustained, the patient is considered to have lupus flare.
  Lupus flare can be further evaluated according to SELENA-SLEDAI Flare Index (SFI).
  Lupus nephritis flare can be further evaluated as flare of proteinuria and flare of nephritis.

SECONDARY OUTCOMES:
The 1-year flare rate of lupus nephritis participants who accept MMF or TAC monotherapy. | 18th~30th month
  If the DORIS (Definition of Remission In SLE) is not sustained, the patient is considered to have lupus flare.
Lupus flare (as assessed by SLEDAI and PGA) in SLE patients during the maintenance period after steroid tapering. | 6th~30th month
The changes of serum activity markers (anti-dsDNA antibody and C3 level) in SLE patients after steroid tapering. | 6th~30th month
Proportion of SLE patients with irreversible organ damage (assessed by SLICC/SDI) after steroid tapering. | 6th~30th month
Changes in carotid intima-media thickness after steroid tapering. | 6th~30th month
Differences in medical charges between steroid tapering and steroid maintenance patients. | 6th~30th month
  Obtain the information by questionnaire.
Differences in health-related quality of life between steroid tapering and steroid maintenance patients. | 6th~30th month
  Evaluate health-related quality of life by Short-Form Six-Dimension (SF-6D) health index. SF-6D includes 6 dimensions: physical functioning, role limitations, social functioning, pain, mental health, and vitality. The minimum total value is 0. The maximum total value is 1. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mengtao Li, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murimi-Worstell IB, Lin DH, Nab H, Kan HJ, Onasanya O, Tierce JC, Wang X, Desta B, Alexander GC, Hammond ER. Association between organ damage and mortality in systemic lupus erythematosus: a systematic review and meta-analysis. BMJ Open. 2020 May 21;10(5):e031850. doi: 10.1136/bmjopen-2019-031850. PMID 32444429
- [Background] Zonana-Nacach A, Barr SG, Magder LS, Petri M. Damage in systemic lupus erythematosus and its association with corticosteroids. Arthritis Rheum. 2000 Aug;43(8):1801-8. doi: 10.1002/1529-0131(200008)43:83.0.CO;2-O. PMID 10943870
- [Background] Fanouriakis A, Kostopoulou M, Alunno A, Aringer M, Bajema I, Boletis JN, Cervera R, Doria A, Gordon C, Govoni M, Houssiau F, Jayne D, Kouloumas M, Kuhn A, Larsen JL, Lerstrom K, Moroni G, Mosca M, Schneider M, Smolen JS, Svenungsson E, Tesar V, Tincani A, Troldborg A, van Vollenhoven R, Wenzel J, Bertsias G, Boumpas DT. 2019 update of the EULAR recommendations for the management of systemic lupus erythematosus. Ann Rheum Dis. 2019 Jun;78(6):736-745. doi: 10.1136/annrheumdis-2019-215089. Epub 2019 Mar 29. PMID 30926722
- [Background] Tani C, Elefante E, Signorini V, Zucchi D, Lorenzoni V, Carli L, Stagnaro C, Ferro F, Mosca M. Glucocorticoid withdrawal in systemic lupus erythematosus: are remission and low disease activity reliable starting points for stopping treatment? A real-life experience. RMD Open. 2019 Jun 11;5(2):e000916. doi: 10.1136/rmdopen-2019-000916. eCollection 2019. PMID 31275608
- [Background] Mathian A, Pha M, Haroche J, Cohen-Aubart F, Hie M, Pineton de Chambrun M, Boutin THD, Miyara M, Gorochov G, Yssel H, Cherin P, Devilliers H, Amoura Z. Withdrawal of low-dose prednisone in SLE patients with a clinically quiescent disease for more than 1 year: a randomised clinical trial. Ann Rheum Dis. 2020 Mar;79(3):339-346. doi: 10.1136/annrheumdis-2019-216303. Epub 2019 Dec 18. PMID 31852672
- [Background] Villarroel MC, Hidalgo M, Jimeno A. Mycophenolate mofetil: An update. Drugs Today (Barc). 2009 Jul;45(7):521-32. doi: 10.1358/dot.2009.45.7.1384878. PMID 19834629
- [Background] Fanouriakis A, Kostopoulou M, Cheema K, Anders HJ, Aringer M, Bajema I, Boletis J, Frangou E, Houssiau FA, Hollis J, Karras A, Marchiori F, Marks SD, Moroni G, Mosca M, Parodis I, Praga M, Schneider M, Smolen JS, Tesar V, Trachana M, van Vollenhoven RF, Voskuyl AE, Teng YKO, van Leew B, Bertsias G, Jayne D, Boumpas DT. 2019 Update of the Joint European League Against Rheumatism and European Renal Association-European Dialysis and Transplant Association (EULAR/ERA-EDTA) recommendations for the management of lupus nephritis. Ann Rheum Dis. 2020 Jun;79(6):713-723. doi: 10.1136/annrheumdis-2020-216924. Epub 2020 Mar 27. PMID 32220834
- [Background] Mok CC. Mycophenolate mofetil for non-renal manifestations of systemic lupus erythematosus: a systematic review. Scand J Rheumatol. 2007 Sep-Oct;36(5):329-37. doi: 10.1080/03009740701607042. PMID 17963161
- [Background] Broen JCA, van Laar JM. Mycophenolate mofetil, azathioprine and tacrolimus: mechanisms in rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):167-178. doi: 10.1038/s41584-020-0374-8. Epub 2020 Feb 13. PMID 32055040
- [Background] Yoon KH. Efficacy and cytokine modulating effects of tacrolimus in systemic lupus erythematosus: a review. J Biomed Biotechnol. 2010;2010:686480. doi: 10.1155/2010/686480. Epub 2010 Jun 28. PMID 20625508
- [Background] Hannah J, Casian A, D'Cruz D. Tacrolimus use in lupus nephritis: A systematic review and meta-analysis. Autoimmun Rev. 2016 Jan;15(1):93-101. doi: 10.1016/j.autrev.2015.09.006. Epub 2015 Sep 30. PMID 26427983
- [Background] Zhang H, Liu Z, Zhou M, Liu Z, Chen J, Xing C, Lin H, Ni Z, Fu P, Liu F, Chen N, He Y, Liu J, Zeng C, Liu Z. Multitarget Therapy for Maintenance Treatment of Lupus Nephritis. J Am Soc Nephrol. 2017 Dec;28(12):3671-3678. doi: 10.1681/ASN.2017030263. Epub 2017 Jul 31. PMID 28760751
- [Background] Peng L, Wang Z, Li M, Wang Y, Xu D, Wang Q, Zhang S, Zhao J, Tian X, Zeng X. Flares in Chinese systemic lupus erythematosus patients: a 6-year follow-up study. Clin Rheumatol. 2017 Dec;36(12):2727-2732. doi: 10.1007/s10067-017-3842-z. Epub 2017 Sep 19. PMID 28929239